CLINICAL TRIAL: NCT03638999
Title: A Prospective, Randomized, Pilot Study of Preoperative Anti-Inflammatory Therapy for Ureteral Stent Symptoms
Brief Title: NSAIDs Stent Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 201804199
Record Dates: First submitted 2018-07-26; First posted 2018-08-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Ureteral Stent Placement; Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Ketorolac; Injections; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in 1:1 ratio to either intervention or control group. Subjects in the intervention group will receive intravenous injection of 1 ml of Ketorlac 30 mg/ml, whereas subjects in the control group will receive 1 ml of 0.9% injectable normal saline, prior to the start of the procedure. Study team, with the exception of the pharmacist, will be blinded to randomization results.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Prior to initiation of study enrollment, envelopes containing study randomization assignments will be created, sequentially numbered, sealed and given to the study pharmacist. Once a patient provides consent and meets study inclusion and exclusion criteria, study pharmacist will be notified of enrollment and will randomize the patient by opening the next subsequent randomization envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention Group - Ketorlac (NSAID) (Active Comparator): Subjects will receive a one-time intravenous injection of 1 ml of Ketorlac 30 mg/ml prior to the start of the ureteroscopic procedure. After consent and during screening visit demographic information, medical/surgical history, and height and weight will be collected. On Day 0 subject will be randomized to NSAID or Saline using inclusion/exclusion criteria and the procedure data will be collected. On Day 1 subject will receive a follow up phone call and complete AUA Symptom Score, USS Questionnaire 1 and USS Questionnaire 2 and any adverse events will be assessed. These questionnaires will again be administered on the day of stent removal and again 1 to 2 months post stent removal.
  Interventions: Drug: Ketorolac Trometamol 30Mg/1mL Injection
- Placebo Group - Normal Saline (Placebo Comparator): Subjects in the control group will receive a one-time 1 ml of 0.9% injectable normal saline prior to the start of the ureteroscopic procedure. After consent and during screening visit demographic information, medical/surgical history, and height and weight will be collected. On Day 0 subject will be randomized to NSAID or Saline using inclusion/exclusion criteria and the procedure data will be collected. On Day 1 subject will receive a follow up phone call and complete AUA Symptom Score, USS Questionnaire 1 and USS Questionnaire 2 and any adverse events will be assessed. These questionnaires will again be administered on the day of stent removal and again 1 to 2 months post stent removal.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketorolac Trometamol 30Mg/1mL Injection — Subjects in the intervention group will receive intravenous injection of 1 ml of Ketorlac 30 mg/ml prior to the start of the ureteroscopic procedure.
  Other Names: Toradol IV/IM
  Arms: Intervention Group - Ketorlac (NSAID)
Drug: Normal saline — Subjects in the control group will receive 1 ml of 0.9% injectable normal saline prior to the start of the ureteroscopic procedure.
  Arms: Placebo Group - Normal Saline

SUMMARY:
This is a pilot study to (1) evaluate the effect of Ketorolac on inflammatory response and its impact on stent related symptoms in patients undergoing stent placement procedure and (2) assess feasibility of recruitment, randomization, assessment procedures and implementation of the study intervention.

DETAILED DESCRIPTION:
Ureteral stent is routinely placed following ureteroscopic procedures to aid in urinary drainage post-operatively. Up to 80% of patients, however, experience stent-related symptoms (SRS) including lower abdominal pain, burning with urination, blood in urine and voiding symptoms affecting activities of their daily living. Intra- and/or post-operative therapeutic options are limited and most are initiated following the ureteral stent placement when the inflammatory process has already begun from ureteral manipulation, further limiting their efficacy. We, therefore, hypothesize that pre-operative intravenous administration of Ketorolac, with its anti-inflammatory and analgesic properties, will reduce the inflammatory process during ureteral manipulation and reduce SRS.

The eligible patients undergoing ureteral stent placement will be randomized 1:1 into either intervention or control group. Subjects in the intervention group will receive intravenous injection of 1 ml of Ketorlac 30 mg/ml, whereas subjects in the control group will receive 1 ml of 0.9% injectable normal saline, prior to the start of the procedure. A panel of plasma inflammatory markers will be drawn and assessed pre- and post-operatively as well as at the time of stent removal as an objective measures for inflammation.

A follow-up telephone call will be made by the nursing staff on post-operative day one to check on patient status and to re-educate the patients to follow the protocol.

To assess SRS, all participants will complete the AUA Symptom Score Questionnaire and the Analog Pain Scale prior to the procedure. On post-operative day 1 and at the time of stent removal (prior to the stent being taken out), participants will complete the USSQ1 and the AUA Symptom Score. At the time of subsequent follow up visit, participants will complete the USSQ2 and AUA Symptom Score.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age and willing and able to provide informed consent
* Patients with renal urolithiasis planning to undergo ureteral stent placement following ureteroscopic manipulation

Exclusion Criteria:

* Patients requiring a bilateral stone procedure.
* Patients on a chronic non-steroidal anti-inflammatory drugs (NSAIDs) including Aspirin defined as any NSAIDs use for more than fifteen days within thirty days prior to the procedure. Exception: use of daily Aspirin 81 mg is allowed.
* Patients on any steroid therapy.
* Patients with prescription anti-inflammatory drugs.
* Patients with gastrointestinal ulcers.
* Patients with ureteral obstruction or stricture unrelated to stone disease.
* Patients with active urinary tract infection as evidence of untreated positive urine culture obtained prior to the procedure (as part of pre-operative testing).
* Patients with preexisting indwelling ureteral stent
* Patients who are pregnant or lactating.
* Patients with renal or liver impairment.
* Patients with concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would render the patient inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Analog Pain Scale, 0 - 10 rating of pain - Stent insertion Day 1 | Stent insertion Day 1
  The Analog Pain Scale is a patient reported scale from 0-10 that will be administered after standard surgical procedure of ureteroscopy with or without laser lithotripsy and/or stone extraction). The Analog Pain Scale uses 0 (zero) to describe no pain and 10 will reference worst pain.
Analog Pain Scale, 0 - 10 rating of pain - Stent removal | Stent removal visit (Approximately 7 to 14 days)
  The Analog Pain Scale is a patient reported scale from 0-10 that will be administered during the stent removal visit. The Analog Pain Scale uses 0 (zero) to describe no pain and 10 will reference worst pain.
Analog Pain Scale, 0 - 10 rating of pain - Follow-up Visit | 1 to 2 months post stent removal
  The Analog Pain Scale is a patient reported scale from 0-10 that will be administered during follow up visit. The Analog Pain Scale uses 0 (zero) to describe no pain and 10 will reference worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Alana Desai, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Assimos D, Krambeck A, Miller NL, Monga M, Murad MH, Nelson CP, Pace KT, Pais VM Jr, Pearle MS, Preminger GM, Razvi H, Shah O, Matlaga BR. Surgical Management of Stones: American Urological Association/Endourological Society Guideline, PART II. J Urol. 2016 Oct;196(4):1161-9. doi: 10.1016/j.juro.2016.05.091. Epub 2016 May 27. PMID 27238615
- [Background] Joshi HB, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG, Barry MJ. Indwelling ureteral stents: evaluation of symptoms, quality of life and utility. J Urol. 2003 Mar;169(3):1065-9; discussion 1069. doi: 10.1097/01.ju.0000048980.33855.90. PMID 12576847
- [Background] Lamb AD, Vowler SL, Johnston R, Dunn N, Wiseman OJ. Meta-analysis showing the beneficial effect of alpha-blockers on ureteric stent discomfort. BJU Int. 2011 Dec;108(11):1894-902. doi: 10.1111/j.1464-410X.2011.10170.x. Epub 2011 Mar 31. PMID 21453351
- [Background] Norris RD, Sur RL, Springhart WP, Marguet CG, Mathias BJ, Pietrow PK, Albala DM, Preminger GM. A prospective, randomized, double-blinded placebo-controlled comparison of extended release oxybutynin versus phenazopyridine for the management of postoperative ureteral stent discomfort. Urology. 2008 May;71(5):792-5. doi: 10.1016/j.urology.2007.11.004. Epub 2008 Mar 12. PMID 18339420
- [Background] De Oliveira GS Jr, Agarwal D, Benzon HT. Perioperative single dose ketorolac to prevent postoperative pain: a meta-analysis of randomized trials. Anesth Analg. 2012 Feb;114(2):424-33. doi: 10.1213/ANE.0b013e3182334d68. Epub 2011 Sep 29. PMID 21965355
- [Background] Elwood CN, Lange D, Nadeau R, Seney S, Summers K, Chew BH, Denstedt JD, Cadieux PA. Novel in vitro model for studying ureteric stent-induced cell injury. BJU Int. 2010 May;105(9):1318-23. doi: 10.1111/j.1464-410X.2009.09001.x. Epub 2009 Nov 3. PMID 19888977
- [Background] Beiko DT, Watterson JD, Knudsen BE, Nott L, Pautler SE, Brock GB, Razvi H, Denstedt JD. Double-blind randomized controlled trial assessing the safety and efficacy of intravesical agents for ureteral stent symptoms after extracorporeal shockwave lithotripsy. J Endourol. 2004 Oct;18(8):723-30. doi: 10.1089/end.2004.18.723. PMID 15659891
- [Background] Krambeck AE, Walsh RS, Denstedt JD, Preminger GM, Li J, Evans JC, Lingeman JE; Lexington Trial Study Group. A novel drug eluting ureteral stent: a prospective, randomized, multicenter clinical trial to evaluate the safety and effectiveness of a ketorolac loaded ureteral stent. J Urol. 2010 Mar;183(3):1037-42. doi: 10.1016/j.juro.2009.11.035. Epub 2010 Jan 21. PMID 20092835